CLINICAL TRIAL: NCT00951886
Title: The Validity of Forced Expiratory Maneuvers in Ataxia Teleangiectasia Studied Longitudinally
Brief Title: The Validity of Forced Expiratory Maneuvers in Ataxia Telangiectasia Studied Longitudinally
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sheba medical Center, Ori Efrati, MD, Principal Investigator, Sheba medical Center
Other Study IDs: SHEBA-08-5418-OE-CTIL
Record Dates: First submitted 2009-08-02; First posted 2009-08-04 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Ataxia Telangiectasia
Keywords: Ataxia Teleangiectasia; Spirometry; Respiratory rare diseases
MeSH Terms: conditions — Ataxia Telangiectasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Rationale: Forced spirometry maneuvers are not routinely performed in patients with Ataxia Telangiectasia (A-T), even though they suffer from respiratory illnesses.

Objectives: To study the feasibility and validity of forced spirometry in A-T patients.

Methods: Patients will perform spirometry during clinical visits. Parameters studied will be technical quality, relation to predicted values, age, pulmonary illness, body mass index, mutational status and mutation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven Ataxia Telangiectasia

Exclusion Criteria:

* inability to perform spirometry

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Ataxia Telangiectasia who are followed and treated in the National A-T center at Safra Children's Hospital, Sheba Medical Center, Ramat-Gan, Israel
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2009-07; Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
spirometry measurements | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Pulmonary Unit, The Edmond and Lily Safra Children's Hospital Chaim Sheba Medical Center, Tel HaShomer, Ramat Gan, Israel